CLINICAL TRIAL: NCT05233189
Title: Personalized Massive Online Open Course After Childhood Cancer: Impact Study START-MOOC2
Brief Title: Personalized Massive Online Open Course After Childhood Cancer
Acronym: START_MOOC2
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire de Saint Etienne (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 21CH173; 2021-A02453-38 (Other: ANSM)
Record Dates: First submitted 2022-02-01; First posted 2022-02-10 (Actual); Last update posted 2025-02-10 (Actual); Status verified 2025-02

CONDITIONS: Long-Term Survivors
Keywords: Long-term follow-up; childhood cancer; massive online open course
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Intervention Model Description: "Cohort multiple randomised controlled trial" design. Patients randomized "no MOOC" group will not be aware of the MOOC. Patients randomized group "with MOOC" will be composed of all former patients who will be offered the MOOC, whether they accept it or not
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- With the MOOC "Childhood cancer, living well, after" (Experimental): Quantify the impact of the MOOC's membership on the CCS knowledge about LTFU adapted to the medical history of patients and measure how this MOOC can improve the LTFU care of each CCS.
  Interventions: Other: MOOC
- Without the MOOC "Childhood cancer, living well, after" (Active Comparator): Quantify the impact of the MOOC's non-membership on the CCS knowledge about LTFU adapted to the medical history of patients and measure how this MOOC can improve the LTFU care of each CCS.
  Interventions: Other: No intervention

INTERVENTIONS:
Other: MOOC — Registrants will be offered a personalized e-education consisting of 3 to 11 modules adapted to the treatment received in childhood by each in the form of a MOOC entitled "Cancer in childhood, living well after" over a total duration of about 3 to 7 weeks of training.
  Arms: With the MOOC "Childhood cancer, living well, after"
Other: No intervention — Patients will be followed up until 18 months only
  Arms: Without the MOOC "Childhood cancer, living well, after"

SUMMARY:
Many studies have shown Childhood Cancer Survivors (CCS) are ill-informed about long-term follow-up (LTFU). Massive open online courses (MOOCs) could easily allow a deployment at an international level and make reliable information available for all CCS, wherever they live. The MOOC team (specialists of LTFU care, communication professionals and CCS associations), bringing together nearly 130 people, designed a MOOC named "Childhood Cancer, Living Well, After" including three modules addressing transversal issues (lifestyle, psychological support, fertility problems) and eight modules covering organ-specific problems.

DETAILED DESCRIPTION:
Detailed data on childhood cancer treatments were used during a study of feasibility in spring 2020 to allocate specific modules to each participant. The aim of the present study is to quantify the impact of this MOOC on the CCS knowledge about LTFU adapted to their own medical history, but also to measure how this MOOC can improve the LTFU care of each CCS.

ELIGIBILITY:
Inclusion Criteria:

* Patient affiliated or entitled to a social security plan,
* Former patient included in the Childhood Cancer Observation Platform (CCOP) for pediatric cancer or leukemia (<15 years of age) between 2000 and 2010 with at least five years free of anticancer treatment
* Availability of computerized and validated treatment data in the Childhood Cancer Observation Platform (CCOP),
* A subject who has received informed information about the study and digitally signed the online express consent for subjects participating in the MOOC, and digitally signed the online express consent to continue for subjects not participating in the MOOC
* A subject who completed an initial COHOPER survey from Childhood Cancer Observation Platform (CCOP) online self-questionnaire
* Subject who has accepted that data collected as part of the COHOPER survey (including french national health data system (SNDS)) may be reused for scientific research purposes and shared with other research teams,

Exclusion Criteria:

* A subject having already been drawn for the START-MOOC1 feasibility study,
* A subject for whom a doubt, validated by the study coordinating physician, persists on the exact treatment received in childhood and does not allow the allocation of specific modules with certainty,
* A subject who has had several cancers and whose anticancer therapies are not all known,
* A subject who has not been treated in one of the participating referral centers,
* Subject having expressed opposition to the french national health data system (SNDS) interrogation following the sending of the information letter or share the data with other research teams,
* Pregnant

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 532 (Estimated)
Dates: Start 2024-04-30 (Actual); Primary Completion 2025-11 (Estimated); Study Completion 2025-11 (Estimated)

PRIMARY OUTCOMES:
Proportions of former patients with overall adherence to their recommended care pathway. | MONTH 18
  The impact of the MOOC will be measured qualitatively by comparing the two groups "with MOOC" and "without MOOC" of the proportions of former patients with an overall adherence to the care pathway recommended to them.

SECONDARY OUTCOMES:
Level of knowledge of former patients on recommended care pathway. | Month 18
  The quiz concerns 3 modules : "Taking care of yourself after childhood cancer," "Feeling good about yourself, feeling good about yourself," and "Fertility: talking about it!". Global score = 300.
  For each of the 8 specific modules assigned in a personalized way according to the former patients, the average score of the corresponding quiz, also presented in the form of a percentage of correct answers.

CONTACTS AND LOCATIONS:
Overall Officials: Claire BERGER, PHD, Principal Investigator — Centre Hospitalier Universitaire de Saint Etienne
Locations (1):
- CHU de SAINT-ETIENNE, Saint-Etienne, France

IPD SHARING:
Plan to Share IPD: No